CLINICAL TRIAL: NCT03785028
Title: Analysis of Electrocorticographic Signals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-0282; Protocol Version 6/18/2019 (Other: UW Madison); A538900 (Other: UW Madison); SMPH\PSYCHIATRY\PSYCHIATRY (Other: UW Madison); 2R01MH095984 (NIH)
Record Dates: First submitted 2018-12-14; First posted 2018-12-24 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: basic science
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Only arm of this basic science study, participants will undergo working memory and attention tasks
  Interventions: Behavioral: working memory and attention

INTERVENTIONS:
Behavioral: working memory and attention — working memory and attention tasks

SUMMARY:
The objectives of this research are to understand how the brain can keep information in mind ("working memory"), and use this information to guide behavior. The two experiments that fall under this study will collect brain signals from epilepsy patients who are having surgery as part of their treatment. More specifically, these signals will be studied from the time while the patient is performing two cognitive tasks.The endpoints are publication of the results from each of the proposed experiments in peer-reviewed journals.

DETAILED DESCRIPTION:
There are 2 separate experiments proposed, both of which use repeated-measures designs.

1: Electrocorticography (ECoG) study of visual working memory. Each trial from the behavioral task will start by presenting subjects with two visual images, one each from two of these three categories: faces, words, and outdoor scenes. They will then be cued as to which one they'll be tested on with a recognition probe, and after the first probe the cuing-probing process is repeated. Patients selected for this study will have depth electrodes implanted in the left medial temporal lobe and/or grids covering left occipital, temporal, and/or parietal cortex, and suitability of a patient's data for the final dataset will require that a minimum of one stimulus category can be decoded from them. (The precise minimum number of trials required cannot be calculated a priori, because this requires knowing the signal-to-noise ratio in a dataset, a property that is highly variable in electrocorticography data.)

2. Electrocorticography of spatial selective attention. Each trial from the behavioral task will start by presenting subjects with a white "+" on a screen, with each arm pointing to a potential target location. During each 92-trial block of trials, only two 180-degree opposing locations will ever be cued, with one arm of the "+" turning yellow and the opposing one turning blue, to indicate with 75% validity the location at which an oriented Gabor patch will appear (5 degrees from fixation; cue color mapping counterbalanced), requiring a speeded "R/L" tilt judgment. Orthogonal to cue-color configuration, half of the trials in each block will begin with presentation of an "x" that will rotate by 45 degrees with an unpredictable lag (.5 sec +/- .3). On these trials, the cue-to-target interval (i.e., from rotation to "+" to color-cue onset) will be 750 msec. On trials that begin with the onset of a "+", cue-to-target interval will vary unpredictably between 650, 750, and 850 msec. Decomposition of alpha-band oscillations (brain waves cycling at roughly 10 times per second) into components associated with each location will be derived by filtering the whole-scalp signal with weights from the inverted encoding model trained to encode the four critical locations.

ELIGIBILITY:
Inclusion Criteria:

* Participants with implanted electrode arrays who are willing to participate and able to cooperate and follow research instructions will be recruited.
* Must be able to read
* Must be able to name objects
* Must be able to articulate thoughts with spoken language

Exclusion Criteria:

* post-operative pain requiring narcotics
* repeated seizures clouding consciousness
* IQ of 85 and below
* post-operative subdural bleeding
* cerebral pathology affecting the cortical regions from which recordings are made
* women who are pregnant, or who think they may be pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2021-02-21 (Actual); Study Completion 2021-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley R Postle, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants undergoing surgery for epilepsy were recruited at UW hospital Neurology clinic in Madison, Wisconsin, from 7/19/19 - 2/27/21.
Groups:
- Experimental Arm: 1 session of a computer-based visual working memory task (~20 minutes total) with concurrent electrocorticography (ECoG) recording.
Period: Overall Study
Arm/Group | Experimental Arm
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental Arm: Participants will undergo working memory and attention tasks
Arm/Group | Experimental Arm
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Measure: Prioritization Cue-related Changes in the Neural Representation of Stimuli Reported as Binary for Prioritized and Unprioritized Item Decodability
Description: This experiment will use a machine learning analysis -- multivariate pattern classification -- to "decode" the brain signals measured by the electrocorticography electrodes. That is, the analysis will determine if the face/word/scene that is being remembered is being represented by these particular brain signals). The primary outcome will be to assess what happens to the neural representation of, say, a face, when the patient is probed that the other stimulus presented on that trial will be tested first - i.e., the analysis will assess the decodability of the two items as a function of their priority for upcoming task demands. Reported here is the categorical performance of Support Vector Machines (SVMs) trained using a 10-fold cross-validation procedure to decode the prioritized and unprioritized memory items (faces, scenes, or words).
Time Frame: Twenty minutes
Population: Data collected from 4 participants, reported here as a group. Three of them completed 5 blocks of 20 trials each, resulting in a total of 100 trials, and one of them completed 4 blocks, 80 trials in total. One participant struggled to perform the task so data were not interpretable.
Measure: Count of Units; unit: group of all participants
Units Other Than Participants: group of all participants
Groups:
- Theta: 3-7 Hz
- Alpha: 8-12 Hz
- Beta: 13-20 Hz
- Gamma: 30-60 Hz (low); 60-200 Hz (high)
Arm/Group | Theta | Alpha | Beta | Gamma
Number analyzed (Participants) | 4 | 4 | 4 | 4
Number analyzed (group of all participants) | 1 | 1 | 1 | 1
group of all participants
  Decoded - Prioritized item | 1 | 1 | 1 | 0
  Not Decoded - Prioritized item | 0 | 0 | 0 | 1
  Decoded - Unprioritized item | 1 | 1 | 0 | 0
  Not decoded - Unprioritized item | 0 | 0 | 1 | 1

2. Primary Outcome: Qualitative Measure: Working Memory Delay Period Phase-amplitude Coupling Reported as Direction (Increase/Decrease) for Region and Stimulus Type
Description: Phase-amplitude coupling (PAC) refers to the synchrony between low frequency oscillations and bursts of high-frequency signal, which is interpreted as a proxy for neuronal firing. The primary outcome measure is whether the level of phase-amplitude coupling associated with a stimulus will change (increase, decrease, change to different frequencies) after that stimulus is prioritized or deprioritized by the cue. Reported here is the direction of PAC between low theta oscillations (6 Hz) and high-gamma bursts (>140 Hz) in binary terms according to whether the PAC increased or decreased for the three stimulus types (faces, scenes, or words) in electrode signals analyzed in different brain regions.
Time Frame: Twenty minutes
Population: Data collected from a single participant, participant had electrodes positioned in each of the target regions to be analyzed to support a within-subject comparison.
Measure: Count of Units; unit: number of electrodes
Units Other Than Participants: number of electrodes
Groups:
- Left Hippocampus; Inferior Temporal Cortex: 1 electrode/contact
- Right Post Temporoparietal: 2 electrodes/contacts were analyzed individually
Arm/Group | Left Hippocampus | Right Post Temporoparietal | Inferior Temporal Cortex
Number analyzed (Participants) | 1 | 1 | 1
Number analyzed (number of electrodes) | 1 | 2 | 1
number of electrodes
  Faces - Decrease | 1 | 1 | 0
  Faces - Increase | 0 | 1 | 1
  Scenes - Decrease | 1 | 0 | 0
  Scenes - Increase | 0 | 2 | 1
  Words - Decrease | 1 | 0 | 1
  Words - Increase | 0 | 2 | 0

3. Primary Outcome: Experiment 3.b. Covert Spatial Attention-related Changes in Phase-amplitude Coupling
Description: Phase-amplitude coupling refers to the synchrony between low frequency oscillations and bursts of high-frequency signal, which is interpreted as a proxy for neuronal firing. The primary outcome measure is whether the level of phase-amplitude coupling in tissue representing a region of space that is irrelevant for an entire block of trials will change in a manner that mirrors the dynamic changes expected for each trial's uncued location, or whether it will be insensitive to shifts of attention that are, by definition, never relevant for that tissue over the course of that block of trials.
Time Frame: Twenty minutes
Population: Experiment was not conducted, so no data available.
Arm/Group | Experimental Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Data collection took ~20 minutes per participant.
Arm/Group | Experimental Arm
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
Study underpowered for meaningful results. Working memory tasks prove challenging for this patient population, leading to unreliable or uninterpretable data. Recruitment challenges related to coverage of data recording, and cognitive ability requirements, are prevalent in this patient population leading to small number of data sets collected and analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT03785028/Prot_SAP_000.pdf